CLINICAL TRIAL: NCT05190497
Title: Effects of Inspiratory Muscle Training on Clinical Predictors of Respiratory Muscle Strength and Lung Function in Burned Patients With Inhalation Injury
Brief Title: Effects of IMT on Pulmonary Functions IN CASES With Inhalation Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Takey Ahmed, Asssociate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IMT in inhalation injury
Record Dates: First submitted 2021-12-11; First posted 2022-01-13 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Inhalation Injury; Pulmonary Function; Respiratory Muscle Strength
Keywords: INSPIRATORT TRAINING -INHALATION INJURY

STUDY DESIGN:
Intervention Model Description: The exercise group received inspiratory muscle training in addition to routine chest physiotherapy (group A).
  The Control group received only routine chest physiotherapy (group B).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): inspiratory muscle training in addition to routine chest physiotherapy in the form of (deep breathing, coughing, and early ambulation)
  Interventions: Device: Exercise group
- control (No Intervention): The Control group received only routine chest physiotherapy

INTERVENTIONS:
Device: Exercise group — Maximal respiratory pressure and reflecting muscles strength were measured by a mouth pressure meter
  Other Names: INSPIRATORY MUSCLE TRAINING
  Arms: intervention group

SUMMARY:
The current study aimed to investigate the effect of inspiratory muscle training (IMT) on pulmonary functions (FEV1and FVC), and respiratory muscle strength in patients with inhalation injury, which may prove to be a promising intervention helping to improve exercise tolerance, relieve dyspnea and suggests an improvement in respiratory muscle function.

DETAILED DESCRIPTION:
Forty male patients suffering from inhalation injury were been included in this study, Participants' ages ranged from 20-35 years old. Patients were selected from the burn department, Om El-Masreen hospital, and randomly assigned into two equal groups.

The exercise group received inspiratory muscle training in addition to routine chest physiotherapy in the form of (deep breathing, coughing, and early ambulation) three times per week for four weeks (group A). The Control group received only routine chest physiotherapy (group B). This study obtained ethical approval by the institutional review board of the Faculty of Physical Therapy - Cairo University, with reference number: P.T.REC/012/003431

ELIGIBILITY:
Inclusion criteria:

* Male patients suffering from inhalation injury.
* Participant age ranged from 20-35 years old.
* All patients had the same medical care.
* Participants have received a good explanation of the treatment and measurement device.
* Treatment was conducted one month after inhalation injury.

Exclusion criteria:

Patients were excluded from this study for any of the following cases such as

* Instability of patient's medical condition.
* Presence of any diseases that could affect the study results.
* Participants having respiratory, cardiac, or neurological diseases that affect pulmonary functions.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
PULMONARY FUNCTION TEST | 3 MONTHS
  Each patient's weight in kilograms, and height in meters were recorded and entered the machine. An individual sat in a chair and inhaled deeply before closing their mouth tightly around the tube. Several exercises were carried out until the patient comprehended and was comfortable with the instruction. The patient inhaled deeply and exhaled as quickly as possible into the spirometer(Morgan Trans Flow Test Vicatest p2 (Kent, ME 87 ED, England).
Respiratory muscles Strength Measurement | 3 MONTHS
  Maximal respiratory pressure and reflecting muscles strength were measured by a mouth pressure meter (Pony FX; COSMED, Rome, Italy) in the sitting position. The highest maximal expiratory pressure (MEP) in cmH2O, and maximal inspiratory pressure (MIP) in cmH2O values in three or more attempts were chosen. Investigators calculated the predicted MEP and MIP values based on age, height, and weight

CONTACTS AND LOCATIONS:
Overall Officials: Maha A El monem, Ass Prof, Study Chair — Cairo University
Locations (1):
- Khaled Takey Ahmed, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
At first study protocol and informed consent
Supporting Information: Study Protocol, SAP, ICF
Time Frame: november 2021 - february 2022
Access Criteria: web address

REFERENCES:
- [Background] Gupta K, Mehrotra M, Kumar P, Gogia AR, Prasad A, Fisher JA. Smoke Inhalation Injury: Etiopathogenesis, Diagnosis, and Management. Indian J Crit Care Med. 2018 Mar;22(3):180-188. doi: 10.4103/ijccm.IJCCM_460_17. PMID 29657376